CLINICAL TRIAL: NCT05885100
Title: Prospective Validation Of The Eleveld TCI Model For Propofol In The Malaysian Obese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN22-140
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Total Intravenous Anaesthesia, Eleveld Model, Obes

STUDY DESIGN:
Intervention Model Description: Patients aged 18 years old and above Body mass index of above 25 kg/m2 Patients Undergoing Elective/emergency surgery in UKMMC with an expected duration of 1 hour
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Obesity class 1 (Experimental)
  Interventions: Drug: Eleveld Model
- Obesity class 2 (Experimental)
  Interventions: Drug: Eleveld Model
- Obesity class 3 (Experimental)
  Interventions: Drug: Eleveld Model

INTERVENTIONS:
Drug: Eleveld Model — Target plasma propofol

SUMMARY:
This is a prospective single blinded randomized trial to validate the 2014 published and widely used Eleveld TCI model which is a universal model suitable for use in all age groups and is suitable for all patients even in the extremes of weight.

This study involves 36 patients who meet the inclusion and exclusion criteria that have been set. Once consent obtained patients will undergo surgery utilizing total intravenous anaesthesia via the target control infusion method and plasma levels of propofol will be sampled sequentially for 1 hour during surgery and analysed to compare the difference between the set and measured level of propofol in plasma. From this data obtained the median absolute prediction error calculated. The secondary goal of this study is to assess the BIS-Propofol correlation in the obese population as well as the hemodynamic stability of this particular model in the obese population.

The data from this study will allow a more targeted anaesthetic approach in the obese population and prevent morbidities in our future practice.

DETAILED DESCRIPTION:
Research question 1. Is the newer Eleveld TCI model for propofol applicable in the Malaysian obese population? 2. What is the bias level measured trough median prediction error (MDAPE) when applied to the Malaysian obese individual? Problem Statement

1. No study done in South East Asian obese population
2. Most studies focus on a group of population which are of Caucasian race with different pheno and genotypes compared with Asian population
3. We aim to validate the claim of the developers of the Eleveld TCI model that the median absolute prediction error of this particular model is approximately 20% in all subtypes of populations focusing on the obese population

INTRODUCTION

Total intravenous anaesthesia (TIVA) the process of induction and mantainence of anaesthesia for patients undergoing surgical procedures without the use of volatile agents. Hypnotic agents and opioids may be utilized to assist in the administration of TIVA. Commonly used agents include the use of propofol and remifentanil combined use mainly due to its positive synergistic effect and its low context-sensitive half time(CSHT). [1] TIVA offer many advantageous properties in contrast to volatile agents which include better recovery profile, less post-operative nausea and vomiting and is more environmentally safe. [1] The goal of TIVA is to ensure adequate depth of anaesthesia and rapid recovery and therefore this combination is ideal to aid in our anaesthetic goal. General infusions and intermittent boluses of these agents may not be ideal as different patient demographics influence the rate of elimination and distribution of drugs in the system [2-3,7], hence targeted control infusions (TCI) were introduced in practice to ensure adequate plasma concentrations for induction and mantainence of anaesthesia.

Since the introduction of the Bristol Model for propofol infusions in 1988, various TCI pumps based on different pharmacokinetic models have been developed through the sequential sampling of blood anaesthetic agent levels of healthy volunteers to allow the formulation of different types of pharmacokinetic models. The most popular and currently used TCI model are the Marsh and the Schneider which administers its infusion based on plasma and effect-site respectively however, both of these models have their limitations as they are only suitable for adult use.[4-5] Besides being only suitable for adults, most of these models are formulated for the non-obese population with a body mass index(BMI) of less than 35 kg/m2 and is unable to provide accurate levels in obese individuals due to the altered pharmacokinetics in this population. Changes in the pharmacokinetics of the obese population may predispose patients to inaccuracies of dosing which may lead to awareness or excessive depth of anaesthesia which may cause adverse effects[5-6]. Until recently in 2014, a general pharmacokinetic model for propofol was formulated and was named the Eleveld model[2-3]. Comparing with previous models developed by utilizing healthy volunteers, Eleveld model was developed by combining pharmacokinetic data from multiple studies involving diverse groups of patients and clinical conditions. This allows the formulation of a single pharmacokinetic model from the aggregated data set which in turn provides better identification of plasma levels. The data available on the open TCI website were taken into consideration and a three compartmental pharmacokinetic model was created using the nonlinear mixed effects modeling software (NONMEM) and was referenced to a 170 cm in height and 70 kg non-obese individual[2,3]. Based on this reference individual, multiple data involving various groups of obese and non-obese patients undergoing TIVA were collected and analyzed through allometric scaling. Mathematical models were formulated to estimate the volume of each compartment and a general use model based on the weight of patients was designed termed the Eleveld TCI Model[2].

The Eleveld model is a multi-compartmental pharmacokinetic model of TCI which applies to a wide range of patients of each sex and weight. This particular model is also suitable for use in elderly, pediatric, lean, and obese populations.[2,3]

OBJECTIVE

This is a prospective study to evaluate and validate the performance index of the Eleveld TCI model for use in the obese population in Malaysia. The recruitment process will be done once approved.

Secondary Objective To determine the hemodynamic stability of the eleveld TCI model and determine the BIS-Propofol correlation of the Eleveld TCI model in the obese population

Hypothesis The median absolute performance error of the Eleveld TCI model in obese individuals is between 20-40%

Null Hypothesis The median absolute performance error of the eleveld TCI model in obese individuals is similar to other models and is unable to provide accurate targeting of propofol level in the obese population

MATERIALS AND METHODS This is an Investigator initiated study done in UKMMC. Informed and written consent will be obtained from subjects by the investigator. All medical devices are deemed safe and approved for use on clinical subjects.

Subjects who are eligible for the study will be identified and if consent is given will be brought into the operating theatre with standard monitoring of at least a 3 lead electrocardiogram, non-invasive blood pressure(NIBP) monitoring and saturation of oxygen (SpO2) probe applied, and induction of anesthesia will commence.

In the operating theatre intravenous access will be established for TIVA. A bispectral index monitoring(BIS) will be attached to ensure and guide the adequate depth of anesthesia and monitored throughout anesthesia maintaining levels of 40-60 whilst titrating the dose of propofol. An arterial line monitoring will be inserted before induction under local anesthesia to assist in blood sampling as well as hemodynamic monitoring intraoperatively. The anesthesia team will include a qualified anesthetist a trained general anesthesia nurse and other staff necessary. The analgesia used in the study is in form of TCI Remifentanil given via a three-way valve valve to ensure continuity.

Induction of anaesthesia will commence by starting the TCI Propofol and Remifentanil utilizing the effect site both at 3-4 mcg/ml and 2 ng/ml respectively and titrating the propofol to desired effect to achieve a BIS reading of 40-60 and unconsciousness to call has been achieved. Once unconsciousness is obtained, remifentanil infusion is increased up to 8 ng/ml if hemodynamics is unaffected and stable prior to intubation, to blunt the sympathetic airway reflexes and adjusted throughout surgery depending on the surgical stimulus. IV rocuronium 0.9 mg/kg will be administered to facilitate endotracheal intubation via the rapid sequence intubation. The TCI propofol is maintained and set to achieve a BIS level of 40-60 throughout procedure.

Blood samples at will be taken following induction. A total of 6 blood samples of 3 ml each will be obtained at intervals of 5,10,20,30,40,60 will be obtained and analysed for propofol concentration via the high performance liquid chromatography method. If there is a recent change of propofol level was done, sampling will be delayed by 3 mins to allow equilibration of blood propofol levels.

Blood samples will be stored in EDTA tubes at room temperature for a maximum of 60 minutes and followed by centrifugation and plasma transferred to cryovials and stored at a temperature of -80 degrees Celsius until analysis.

Sample size calculation

The alpha value is set at 0.05 and 80% power of the study. The sample size is calculated based on Vellinga et al study which showed <20% bias in propofol level of Eleveld model in obese adults citation. The calculation is as follows citation (Yamane) : n = Z 2 ϭ 2 /e 2 where ϭ 2 = variance, e = level of precision, and Z = 1.96 at α 0.05 and power study at 80%. n = (1.96) 2 (2.0) 2 /0.5 2 n = 32 For this study which includes a 10% dropout rate, the total sample size would be 36 subjects.

Statistical test:

All data analysis will be performed using SPSS for Windows version 25.0 (IBM Corp, Armonk, NY, USA). Results will be presented as mean ± standard deviation, median (interquartile range), or frequency (percentages) where appropriate. For between-group analysis, an independent t-test will be used and if the data is skewed, the Mann-Whitney U test will be applied. The qualitative data analysis will be done using the Chi-square test or Fisher exact test as appropriate. A p-value <0.05 will be considered statistically significant.

REFERENCES

1. Z Al-Rifai, MBChB (Hons) MPharm (Hons) FRCA, D Mulvey, BSc (Hons) MBBS MD FRCA, Principles of total intravenous anesthesia: practical aspects of using total intravenous anesthesia, BJA Education, Volume 16, Issue 8, August 2016, Pages 276-280, https://doi.org/10.1093/bjaed/mkv074
2. Eleveld, Douglas J. PhD*; Proost, Johannes H. PhD*; Cortínez, Luis I. MD†; Absalom, Anthony R. MD*; Struys, Michel M. R. F. MD*‡. A General Purpose Pharmacokinetic Model for Propofol. Anesthesia & Analgesia: June 2014 - Volume 118 - Issue 6 - p 1221-1237 DOI: 10.1213/ANE.0000000000000165
3. Vellinga, R., Hannivoort, L. N., Introna, M., Touw, D. J., Absalom, A. R., Eleveld, D. J., & Struys, M. M. R. F. (2021). Prospective clinical validation of the Eleveld propofol pharmacokinetic-pharmacodynamic model in general anesthesia. British Journal of Anaesthesia, 126(2), 386-394. https://doi.org/10.1016/j.bja.2020.10.027
4. Schnider TW, Minto CF, Gambus PL, Andresen C, Goodale DB, Shafer SL, Youngs EJ. The influence of method of administration and covariates on the pharmacokinetics of propofol in adult volunteers. Anesthesiology. 1998 May;88(5):1170-82. DOI: 10.1097/00000542-199805000-00006. PMID: 9605675.
5. Marsh B, White M, Morton N, Kenny GN. Pharmacokinetic model driven infusion of propofol in children. Br J Anaesth 1991;67:41-8
6. Cortínez LI, De la Fuente N, Eleveld DJ, Oliveros A, Crovari F, Sepulveda P, Ibacache M, Solari S. Performance of propofol target-controlled infusion models in the obese: pharmacokinetic and pharmacodynamic analysis. Anesth Analg. 2014 Aug;119(2):302-310. DOI: 10.1213/ANE.0000000000000317. PMID: 24977639.
7. van Kralingen S, Diepstraten J, Peeters MY, Deneer VH, van Ramshorst B, Wiezer RJ, van Dongen EP, Danhof M, Knibbe CA. Population pharmacokinetics and pharmacodynamics of propofol in morbidly obese patients. Clin Pharmacokinet 2011;50:739-50
8. Absalom AR, Mani V, De Smet T, Struys MM. Pharmacokinetic models for propofol-defining and illuminating the devil in the detail. Br J Anaesth 2009;103:26-37
9. van Kralingen S, Diepstraten J, Peeters MY, Deneer VH, van Ramshorst B, Wiezer RJ, van Dongen EP, Danhof M, Knibbe CA. Population pharmacokinetics and pharmacodynamics of propofol in morbidly obese patients. Clin Pharmacokinet 2011;50:739-50
10. Yamane T. Statistics, An Introductory Analysis. 2nd ed. New York: Harper and Row, 19

    .

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years old and above Body mass index of above 25 kg/m2 Patients Undergoing Elective/emergency surgery in UKMMC with an expected duration of 1 hour

Exclusion Criteria:

Patients receiving sedative pre anaesthetic medications from the benzodiazepine group of medications Patients who are in overt sepsis with hemodynamic compromise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
evaluate and validate the performance index of the Eleveld TCI model for use in the obese population in Malaysia | 1.5 years
  Plasma level of Eleveld model

IPD SHARING:
Plan to Share IPD: No